CLINICAL TRIAL: NCT03032601
Title: Physiological Effects of N-Acetyl Cysteine in Patients With Multiple Sclerosis
Acronym: MSNAC
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Principal Investigator, Andrew Newberg, Professor, Department of Integrative Medicine and Nutritional Sciences; Professor, Department of Radiology, Thomas Jefferson University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: 16D.672
Record Dates: First submitted 2017-01-19; First posted 2017-01-26 (Estimated); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Multiple Sclerosis
Keywords: MS (Multiple Sclerosis); Acute Fulminating; Sclerosis; 18F-2-fluoro-2-deoxy-D-glucose fluorodeoxyglucose; 18F Fluorodeoxyglucose 2-Fluoro-2-deoxy-D-glucose (18 FDG); Fludeoxyglucose F 18; Fluorine-18-fluorodeoxyglucose; Positron Emission Tomography (PET); Magnetic Resonance Imaging (MRI); PET MRI; Acetylcysteine; N-acetyl cysteine (NAC); Oral supplements; functional magnetic resonance imaging (fMRI); FDG positron emission tomography (FDG PET)
MeSH Terms: conditions — Multiple Sclerosis; Sclerosis | interventions — Acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- N-acetyl Cysteine Cohort (Active Comparator): Intravenous N-acetyl Cysteine - 50mg in 200ml of D5W over one hour 1 x per week Oral N-acetyl Cysteine - 1 500mg tablet 2 x per day (on days IV N-acetyl cysteine is not administered)
  Interventions: Dietary Supplement: N-acetyl Cysteine
- Control Cohort (No Intervention): Standard of Care Treatment

INTERVENTIONS:
Dietary Supplement: N-acetyl Cysteine — The study consists of two arms. The first arm of this study will receive intravenous and oral NAC, a strong antioxidant that increases brain glutathione, which may be beneficial in MS. NAC, is the N-acetyl derivative of the naturally occurring amino acid, L-cysteine. It is a common over-the-counter supplement that is also available as an injectable pharmaceutical that protects the liver in cases of acetaminophen overdose. It has the potential to reduce markers of oxidative damage, protect against cell death, and to increase glutathione in blood, which might be useful in preventing oxidative damage in MS patients. The second arm will be a waitlist control receiving standard MS care. It should be noted that both arms will receive standard of care while enrolled into the study.
  Arms: N-acetyl Cysteine Cohort

SUMMARY:
Multiple Sclerosis (MS) is a disease in which the myelin surrounding the nerve cells is damaged which affects functioning. MS usually is treated with medications designed to reduce the occurrence of future MS events. Evidence suggests that an important part of the disease process is damage to the myelin and brain caused by too much oxygen (sometimes called oxidative stress) or too much inflammation (or swelling).

The overall goal of this study will be to determine whether N-acetyl cysteine (NAC) will help to support cerebral function in patients with Multiple Sclerosis (MS). This positron emission tomography magnetic resonance imaging (PET-MRI) study will utilize 18F-2-fluoro-2-deoxy-D-glucose fluorodeoxyglucose positron emission tomography FDG PET to measure cerebral metabolism, along with MRI analysis, to measure metabolism and structural effects of NAC in patients with MS.

DETAILED DESCRIPTION:
The original protocol consisted of two arms. The first arm of this study will receive intravenous and oral NAC, a strong antioxidant that increases brain glutathione. NAC, is the N-acetyl derivative of the naturally occurring amino acid, L-cysteine. It is a common over-the-counter supplement that is also available as an injectable pharmaceutical that protects the liver in cases of acetaminophen overdose. Laboratory studies have displayed some benefits to use of NAC. It has the potential to reduce markers of oxidative damage, protect against cell death, and to increase glutathione in blood, which might be useful in preventing oxidative damage in MS patients. The second arm will be a waitlist control receiving standard MS care. It should be noted that both arms will receive standard of care treatment for MS while enrolled in the study.

We amended this protocol to increase the enrollment with an additional 30 participants: 15 in a waitlist group and 15 will receive NAC. Subjects be randomized to either receive NAC or be placed in a waitlist control group. Those patients receiving NAC would receive a combination of IV and oral NAC for 4 months. We may obtain NAC serum measures that require a blood draw at three time points, one at scanning before receiving any NAC, one after the first infusion dose of NAC before the second dose, and another one at the last scan and the last dose of NAC.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of relapsing remitting MS or progressive MS who do not plan to start a medication during the study, or on stable disease modifying medication (interferon, glatiramer, dimethyl fumarate, teriflunomide).
* Age 18 years old to no upper limit
* Physically independent, ambulatory
* Women of childbearing potential will confirm a negative pregnancy test and must practice effective contraception during the period of pilot study. In addition, male subjects who have a partner of childbearing age should practice effective contraception.
* Participants must be able to complete study procedures in the greater Philadelphia area.

Exclusion Criteria:

* Patients are excluded who have received treatment with intravenous steroids within the past 90 days for reasons other than MS
* Previous brain surgery that would interfere with determination of cerebral metabolism or structure on the FDG PET-MRI.
* Score on Mini-Mental Status examination of 20 or lower.
* Wheelchair-bound or bed-ridden, non-ambulatory.
* Intracranial abnormalities that may complicate interpretation of the brain scans (e.g., stroke, tumor, vascular abnormality affecting the target area).
* History of head trauma with loss of consciousness > 48 hours.
* History of asthma requiring daily medications for adequate management.
* Any medical disorder or physical condition that could reasonably be expected to interfere with the assessment of MS symptoms, or with any of the study assessments including the PET-MRI imaging.
* Patients with evidence of a significant psychiatric disorder by history/examination that would prevent completion of the study will not be allowed to participate.
* Patients with current alcohol or drug abuse
* Pregnant or lactating women.
* Enrollment in active clinical trial/ experimental therapy within the prior 30 days.
* Pending surgery during the course of the study.
* Patients taking medications that might interact with NAC involved in this study will be evaluated on a case by case basis by the PI or study physician. These medications include: Medications for high blood pressure; Medications that slow blood clotting; Medications for diabetes; Nitroglycerin.
* Patients with history of pulmonary hypertension.
* Any neurological, psychiatric, or medical condition that might affect the distribution of the radiopharmaceutical in the body or brain (as determined by Investigator)
* Currently using medications that might alter the distribution of radiopharmaceuticals in - -the body or brain (as determined by Investigator)
* Patient exceeds the weight limit of the table
* Claustrophobia that would prevent completion of imaging studies
* Glucose level that would interfere with the FDG PET scan
* Any additional contraindications for MRI; Has metallic objects (e.g., pacemakers) in the body

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2017-01-05 (Actual); Primary Completion 2027-07-08 (Estimated); Study Completion 2027-07-08 (Estimated)

PRIMARY OUTCOMES:
Changes in the metabolic activity in the brain, and improved parameters with regard to the inflammation associated with the active lesions based on both MRI and PET findings. | Baseline and 60 ± 30 days
  The goal would be to find a shorter duration of active lesions, reduced impact of the lesions on metabolic activity in the brain, and improved parameters with regard to the inflammation associated with the active lesions based on both MRI and PET findings. Changes on the PET and MRI scans would be correlated with changes in clinical findings and quality of life measures.

SECONDARY OUTCOMES:
Mini-Mental Status examination (MMSE) | Determine eligibility
  Questionnaire used to determine eligibility and cognitive function. (exclusion from study if score is 20 or lower)
Multiple Sclerosis Quality of Life Inventory (MSQLI) | Baseline and 60 ± 30 days
  Participants in the intervention and waitlist (standard of care) group will be asked to complete the full MSQLI which includes the following 10 scales - SF-36, MFIS, PES, BLCS, BWCS, IVIS, PDQ, MHI, MSSS, and SSS-W. The scales will be conducted at baseline and 60 ± 30 days concurrent to baseline and post scans.
Health Status Questionnaire (SF-36) standard form | Baseline and 60 ± 30 days
  Questionnaire from Multiple Sclerosis Quality of Life Inventory that evaluates the quality of life for those diagnosed with Multiple Sclerosis (MS). Will be used to determine improvements in MS symptoms.
Modified Fatigue Impact Scale (MFIS) standard form | Baseline and 60 ± 30 days
  Questionnaire from Multiple Sclerosis Quality of Life Inventory that evaluates the quality of life for those diagnosed with Multiple Sclerosis (MS). Will be used to determine improvements in MS symptoms.
MOS Pain Effects Scale (PES) | Baseline and 60 ± 30 days
  Questionnaire from Multiple Sclerosis Quality of Life Inventory that evaluates the quality of life for those diagnosed with Multiple Sclerosis (MS). Will be used to determine improvements in MS symptoms.
Bladder Control Scale (BLCS) | Baseline and 60 ± 30 days
  Questionnaire from Multiple Sclerosis Quality of Life Inventory that evaluates the quality of life for those diagnosed with Multiple Sclerosis (MS). Will be used to determine improvements in MS symptoms.
Bowel Control Scale (BWCS) | Baseline and 60 ± 30 days
  Questionnaire from Multiple Sclerosis Quality of Life Inventory that evaluates the quality of life for those diagnosed with Multiple Sclerosis (MS). Will be used to determine improvements in MS symptoms.
Impact of Visual Impairment Scale (IVIS) | Baseline and 60 ± 30 days
  Questionnaire from Multiple Sclerosis Quality of Life Inventory that evaluates the quality of life for those diagnosed with Multiple Sclerosis (MS). Will be used to determine improvements in MS symptoms.
Perceived Deficits Questionnaire (PDQ) standard form | Baseline and 60 ± 30 days
  Questionnaire from Multiple Sclerosis Quality of Life Inventory that evaluates the quality of life for those diagnosed with Multiple Sclerosis (MS). Will be used to determine improvements in MS symptoms.
Mental Health Inventory (MHI) standard form | Baseline and 60 ± 30 days
  Questionnaire from Multiple Sclerosis Quality of Life Inventory that evaluates the quality of life for those diagnosed with Multiple Sclerosis (MS). Will be used to determine improvements in MS symptoms.
MOS Modified Social Support Survey (MSSS) standard form | Baseline and 60 ± 30 days
  Questionnaire from Multiple Sclerosis Quality of Life Inventory that evaluates the quality of life for those diagnosed with Multiple Sclerosis (MS). Will be used to determine improvements in MS symptoms.
Sexual Satisfaction Scale (SSS) | Baseline and 60 ± 30 days
  Questionnaire from Multiple Sclerosis Quality of Life Inventory that evaluates the quality of life for those diagnosed with Multiple Sclerosis (MS). Will be used to determine improvements in MS symptoms.
Kurtzke Expanded Disability Status Scale (EDSS) | Baseline and 60 ± 30 days
  Used to measure neurological impairment in those diagnosed with Multiple Sclerosis on a scale of 0 to 10. Will be used to determine improvements in MS symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel A Monti, MD, MBA, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Result] Shahrampour S, Heholt J, Wang A, Vedaei F, Mohamed FB, Alizadeh M, Wang Z, Zabrecky G, Wintering N, Bazzan AJ, Leist TP, Monti DA, Newberg AB. N-acetyl cysteine administration affects cerebral blood flow as measured by arterial spin labeling MRI in patients with multiple sclerosis. Heliyon. 2021 Jul 16;7(7):e07615. doi: 10.1016/j.heliyon.2021.e07615. eCollection 2021 Jul. PMID 34377857

DOCUMENTS (1):
  • Informed Consent Form (2021-10-04): https://cdn.clinicaltrials.gov/large-docs/01/NCT03032601/ICF_003.pdf